CLINICAL TRIAL: NCT04025047
Title: A Multi-center Registry Study: The Complications After Women Having Pelvic Reconstruction Surgery With Trans-vaginal Mesh
Brief Title: A Multi-center Registry Study: The Follow-up the Complications for Trans-vaginal Mesh Surgery
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Qilu Hospital of Shandong University (Other); The First Affiliated Hospital of Nanchang University (Other); Jiangxi Maternal and Child Health Hospital (Other); Fuzhou General Hospital (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Affiliated Wuhu Clinical College of Nantong University (Unknown); The Second Hospital of Anhui Medical University (Other); Renmin Hospital of Wuhan University (Other); Second Xiangya Hospital of Central South University (Other); Changsha Hospital for Maternal and Child Health Care (Other); The Third Xiangya Hospital of Central South University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Shenzhen People's Hospital (Other); Fourth Medical Center of PLA General Hospital (Other); Beijing Chao Yang Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); Second Hospital of Jilin University (Other); Shengjing Hospital (Other); Yantai Yuhuangding Hospital (Other); Shanxi Coal Center Hospital (Unknown); Mianyang Central Hospital (Other); West China Second University Hospital (Other); Chongqing Medical Center for Women and Children (Other); Southwest Hospital, China (Other); Shaanxi Provincial People's Hospital (Other); First Affiliated Hospital of Xinjiang Medical University (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Dalian Maternity and Child Care Hospital (Other); Henan Provincial People's Hospital (Other); Shanghai 10th People's Hospital (Other); Shanghai First Maternity and Infant Hospital (Other); Nanjing Maternity and Child Health Care Hospital (Other); Affiliated Renhe Hospital of China Three Gorges University, China (Unknown); Guizhou Provincial People's Hospital (Other); The First Affiliated Hospital of the Medical College, Shihezi University，China (Unknown); Yangpu District Central Hospital Affiliated to Tongji University (Other); Wuhan Central Hospital (Other)
Responsible Party: Principal Investigator, zhulan, MD, the Chief of General Gynecology Center, the Department of Obstetrics & Gynecology, Peking Union Medical College Hospital
Other Study IDs: JS-1979
Record Dates: First submitted 2019-07-17; First posted 2019-07-18 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Pelvic Organ Prolapse
Keywords: trans-vaginal mesh; pelvic reconstruction surgery; complications; the CTS(category-time-site) coding system
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transvaginal mesh: Patients who undergo pelvic reconstruction surgery using trans-vaginal mesh (commercial mesh kits or self-cut synthesized mesh).

SUMMARY:
This is a multi-center, prospective, observational, hospital-based registry of pelvic organ prolapse(POP) patients who having trans-vaginal mesh implantation with 12 month and 36 month follow-up.To investigate the incidence of postoperative complications according to the International Urogynecological Association/International Continence Society (IUGA/ICS) complication classification system(the Category- Time-Site(CTS) coding).

DETAILED DESCRIPTION:
Patients who undergo pelvic floor reconstructive surgery with trans-vaginal mesh for the cure of pelvic organ prolapse (POP) between June 2019 and December 2022 from 41 centers across the country are going to be prospectively collected. The study is designed to report the clinical data，outcomes and complications of transvaginal mesh surgery in China. The information gathered will identify the incidence rate of complications, especially mesh exposure/erosion, in Chinese women and whether published, professional guidelines on POP surgical treatment as well as mesh complications management are being applied appropriately. Findings from this registry may help in knowing the current status of transvaginal mesh use in China as well as identify issues that may affect the surgical outcome and complications occurrence. Based on the registry study, clinical practice on the management of transvaginal mesh implantation including selection patients, pre- and post-operative evaluation and complications surgical database will be established.

The follow-up process starts after patients have completed the operation; thus, our study does not affect patients' choice of surgical method.

ELIGIBILITY:
Inclusion Criteria:

1） Patients who undergo the pelvic reconstruction surgery with trans-vaginal mesh; 2) Patient is mentally able to understand the nature, aims, or possible consequences of the clinical investigation; 3）Willing to participate in 36 months of longitudinal follow-up and able to provide written informed consent. Willing to provide an email address and complete questionnaires on we-chat, either in clinic or elsewhere when they have access to the internet.

Exclusion Criteria:

* 1) Currently pregnant at enrollment;
* 2) Physically or mentally unable to participate in up to 36 months of follow-up;
* 3) Desires other surgical management of POP other than trans-vaginal mesh.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who prefer to undertake pelvic reconstruction surgery with trans-vaginal mesh for 1) a newly diagnosed severe POP: at least stage III (ICS-classification according to POP-Q system) in one or more compartments; 2) The failure or recurrence after pelvic floor reconstruction with native-tissue(symptomatic II and above).
Sampling Method: Probability Sample
Enrollment: 4147 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of complications | 12 months postoperatively
  Postoperative follow-up and record the occurrence of complications according to the International Urogynecological Association-International Continence Society（IUGA-ICS）Complication Classification Coding(Category-Time-Site coding system).
The incidence rate of complications | 36 months postoperatively
  Postoperative follow-up and record the occurrence of complications according to the International Urogynecological Association-International Continence Society（IUGA-ICS）Complication Classification Coding(Category-Time-Site coding system).

SECONDARY OUTCOMES:
Anatomical cure rate in treated compartment of pelvic reconstructive surgery with trans-vaginal mesh | 6 weeks, 3 months and each year, up to 3-year postoperatively
  The percentage of patients who reach the anatomical success criteria at each time point（6 weeks, 3 months and each year, up to 3-year postoperatively）.The anatomical success is defined by a composite outcome that includes absence of vaginal bulge symptoms, absence of vaginal descent beyond the hymen and the absence of retreatment.
Change from preoperative scores of POP-Q(Pelvic organ prolapse quantitation) at each follow-up | Preoperatively; At 6weeks, 3 months, 1 year and assessed up to 3 year postoperatively
  POP-Q is used for evaluation the severity(staging) of prolapse by pelvic examination preoperatively and postoperatively. The score is reported in cm. The changes from baseline scores at 6 weeks, 3 months, 1 year and up to 3 years postoperatively are respectively compared.
Patient global impression of improvement (PGI-I) | At 6weeks, 3 months, 1 year and assessed up to 3 year postoperatively
  The Chinese-version validated questionnaire PGI-I is used for assessing patients' subjective satisfaction to the pelvic floor reconstructions surgery.
  The PGI-I score ranges from 0~7.
Changes in Pelvic Floor Distress Inventory-20 (PFDI-20) scores | Preoperatively; At 1 year and 3 year postoperatively
  The Chinese-version validated questionnaire Pelvic Floor Distress Inventory-short Form 20 scores [PFDI-20] is to evaluate the impact on pelvic floor function.
Changes in Pelvic Floor Impact Questionnaire-7（PFIQ-7）scores | Preoperatively; At 1 year and 3 year postoperatively
  The Chinese-version validated questionnaire Pelvic Floor Impact Questionnaire-7 [PFIQ-7] is to evaluate the impact on quality of life.
Changes in sexual function and measured by the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire（PISQ-12）scores | Preoperatively; At 1 year and 3 year postoperatively
  The Chinese-version validated questionnaire Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire scores （PISQ-12） is to evaluate the impact on sexual function.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, MD, Principal Investigator — Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences, Beijing, Beijing Municipality, China